CLINICAL TRIAL: NCT07289841
Title: Integration of Ostomy Management Skills Discharge Checklist Into Patient Education and Its Effect on Stoma Adaptation and Quality of Life
Brief Title: Discharge Checklist for Stoma Management Skills
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neslihan Özcanarslan (Other)
Responsible Party: Sponsor-Investigator, Neslihan Özcanarslan, Asst.Prof., Toros University
Organization: Toros University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22.06.2022/129
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Over 18 Years Old
Keywords: Skills Discharge Checklist; Adaptation; Discharge; Ostomy; Quality of life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group that used the Stoma Management Skills Discharge Checklist. (Experimental): The Stoma Management Skills Discharge Checklist will be used during discharge.
  Interventions: Other: Stoma Management Skills Discharge Checklist used
- The group that follows the standard discharge process (No Intervention): Discharge checklist will not be applied, it will be in the standard discharge process

INTERVENTIONS:
Other: Stoma Management Skills Discharge Checklist used — It is seen that there is no structured discharge checklist that systematically evaluates the knowledge and skill levels of stoma patients during the discharge process and there are no comprehensive studies addressing the impact of such a list on stoma adaptation and quality of life.
  Arms: The group that used the Stoma Management Skills Discharge Checklist.

SUMMARY:
The aim of this study was to develop an Ostomy Management Skills Discharge Checklist and to prospectively compare individuals who received this list with those who received standard discharge training to monitor its impact on ostomy compliance and quality of life. The study hypotheses were: The developed Stoma Management Skills Discharge Checklist is more effective than standard discharge training in improving ostomy compliance in individuals with stoma.

H1: It is more effective in improving the quality of life in individuals with stoma.

DETAILED DESCRIPTION:
This is a quasi-experimental, prospective study to be conducted between December 2025 and March 2026. An analytical approach will be employed. As part of the study, an Ostomy Management Skills Discharge Checklist will be developed, and individuals who received this list will be prospectively compared with those who received standard discharge training to monitor their adaptation to ostomy and their impact on quality of life.This study will be conducted with patients who underwent new intestinal stomas in the General Surgery, Gastroenterology Surgery, and Surgical Oncology departments of Mersin City Training and Research Hospital. Patients will be selected using the purposive sampling method among those who underwent new stomas (colostomies or ileostomies) after surgery. The sample size was calculated based on data from a pilot study with 10 patients using r = 1 (equal sample size for both groups), α = 5%, and 90% power. The sample size was calculated using the formula N = α(Zα/2 + Z1-β)² (r + 1) / r d² (N = (1 + 1) × (1.96 + 0.84)² × 2 × (1.2)² / [1 × (1.6 - 1.4)²]). As a result of the calculation, 32 patients per group were determined for 90% power. A total of 80 patients with new ostomies were included in the study. 40 of these patients will form Group 1, which will be followed with the standard discharge process, and the other 40 will form Group 2, whose discharge is planned based on the Stoma Management Skills Discharge Checklist.

The study provides all patients with the same discharge education. Group 1 receives standard education without a checklist, while Group 2 is evaluated with the Stoma Management Skills Discharge Checklist to objectively assess readiness for discharge. Patients must reach a sufficient level in all checklist steps, and any missing skills are re-taught individually. About one month after discharge, both groups are assessed for ostomy adaptation and quality of life. Data are collected by the surgical unit nurse responsible for ostomy patients through 15-20-minute face-to-face interviews in a quiet room.

Data will be analyzed using IBM SPSS Statistics 22. Frequencies (number, percentage) will be used for categorical variables, and descriptive statistics (mean, standard deviation) for numerical variables. Normality of numerical variables will be assessed through skewness and kurtosis values; values within ±1.5 will be considered normally distributed, therefore parametric tests will be applied. Relationships between two independent categorical variables will be evaluated with the Chi-Square test, and Fisher's Exact test will be used when Chi-Square assumptions are not met. A significance level of 0.05 will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients with a new stoma
* Admitted to General Surgery, Gastrointestinal Surgery, or Surgical Oncology departments
* Discharged with only a stoma
* Without comorbidities
* Alive after surgery
* Able to independently manage their stoma care

Exclusion Criteria:

* Visual impairments (e.g., partial blindness, advanced cataracts)
* Physical impairments (e.g., tremors, Parkinson's disease, stroke)
* Intellectual disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Descriptive characteristics form | 12 weeks
  This form includes 10 questions covering age, gender, marital status, education level, social security, occupation, the clinic where the patient was hospitalized, whether the surgery was emergency or elective, and the type of ostomy.

SECONDARY OUTCOMES:
Ostomy Adaptation Scale (OAS) | 12 weeks
  Ostomy Adaptation Scale (OAS): The Stoma Adaptation Scale (OAS23) is a 23-item self-assessment scale with a Cronbach's alpha coefficient of 0.874, developed to evaluate the level of adaptation to a stoma in individuals with stomas. The scale consists of four sub-sections: acceptance (items 1, 3, 4, 6, 9, 14, 15, 19, 23), anxiety/worry (items 12, 13, 17, 20, 21), anger (items 2 and 10), and social adjustment (items 5, 7, 8, 11). Additionally, three items (16, 18, and 22) do not belong to any sub-section. Each item on this scale is evaluated on a 5-point Likert scale (0-4 points: Strongly agree, Agree, Undecided, Disagree, Strongly disagree). The scale has a minimum score of 0 and a maximum score of 92, with higher scores indicating better overall balance. Twelve items (2, 5, 7, 8, 10, 11, 12, 13, 16, 17, 18, and 21) are reverse-scored due to negative statements.
Stoma Quality of Life Scale (SQLS) | 12 weeks
  Developed in 2006, the 21-item SQLS assesses the quality of life of individuals with ostomies. The first two items measure overall life satisfaction, scored from 0 (complete dissatisfaction) to 100 (complete satisfaction). The remaining items are divided into three sub-dimensions: work/social life (6 items), sexuality/body image (5 items), and stoma function (6 items). The scale also includes one item related to economic status and skin irritation, which are not part of any sub-dimension. Except for the first two items, the remaining 19 items in the scale are in a 5-point Likert format (1: never, 2: rarely, 3: sometimes, 4: often, and 5: always). The Turkish adaptation of the scale was carried out by Karadağ et al. in 2011. Confirmatory Factor Analysis (CFA) fit indices of the original scale, consisting of five sub-dimensions and 19 items, showed poor model fit. In conclusion, point 14 (I have concerns about access to stoma care products)

IPD SHARING:
Plan to Share IPD: No